CLINICAL TRIAL: NCT06761729
Title: An Exploratory Study for Evaluating the Efficacy, Safety and Tolerability of JT821 in the Intervention of Behavioral Variant Frontotemporal Dementia
Brief Title: The Ketogenic Diet in the Treatment of Behavioral Variant Frontotemporal Dementia
Acronym: JT821
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XWYY-bvFTD-01
Record Dates: First submitted 2024-12-24; First posted 2025-01-07 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Behavioral Variant Frontotemporal Dementia
MeSH Terms: interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Single Group Assignment,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic diet (Experimental): The subjects initially enter the screening phase (≤ 2 weeks); they undergo the titration period (1 week), gradually titrating to the maximum dose stipulated in the protocol or the maximum tolerable dose for the subject; during the treatment period (12 weeks), but if intolerance emerges during the treatment, the subject can revert to the previous tolerated dose for continued treatment.
  The dosage was titrated incrementally until reaching the maximum daily dose of 30g * 3 meals a day as stipulated in the protocol or the maximum tolerable daily dose for the subject. After entering the treatment period (from week 2 to week 13), this dose was maintained for 12 weeks.
  Interventions: Dietary Supplement: Ketogenic diet

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — Ketogenic diet

SUMMARY:
This study is an exploratory clinical research on the use of JT821 (a ketogenic diet formulation) for the treatment of patients with behavioral variant frontotemporal dementia (bvFTD), aiming to evaluate the effectiveness, safety, and tolerability of JT821 in the intervention of bvFTD.

The ketogenic diet (KD) is a low-carbohydrate, adequate protein and high-fat diet. KD was shown to be effective in treating different neurodegenerative diseases.

DETAILED DESCRIPTION:
This is an exploratory clinical research planned to include 20 subjects diagnosed with behavioral variant frontotemporal dementia (bvFTD). The primary aim of the study is to evaluate the tolerability, efficacy, and safety of JT821 in the treatment of bvFTD.

All subjects will undergo a 1-week product titration period before entering a 12 week treatment period.

Efficacy assessments will be conducted at week 4 and week 12 during the treatment period, utilizing the Montreal Cognitive Assessment (MoCA), the Mini-Mental State Examination (MMSE), and the Clinical Dementia Rating (CDR) scale to assesses the overall cognitive function of the subjects. Additionally, the Frontal Assessment Battery (FAB) will evaluate the executive functions of the frontal lobes; the Neuropsychiatric Inventory (NPI) and the Frontal Behavioral Inventory (FBI) assess the neuropsychiatric and behavioral symptoms of patients; the Boston Naming Test (BNT) and the Verbal Fluency Test (VFT) assess language functions.

Safety evaluation will include the vital signs, laboratory tests (fasting blood glucose, blood ketone levels (β-hydroxybutyrate), urinalysis, complete blood count, fasting lipid profile, liver and kidney function), as well as the recording of any adverse events.

Subjects may withdraw from the study at any time. If subjects experience a serious adverse event, become pregnant, are lost to follow-up, show poor adherence, or if the subject or their legal guardian actively requests to withdraw or retracts informed consent, they may be withdrawn based on the investigator's determination. The sponsor reserves the right to terminate the study at any time for special reasons (such as major safety concerns, force majeure, etc.).

A safety follow-up will be conducted two weeks after the termination of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between the ages of 45 - 70;
2. Meetting the diagnostic criteria for "probable bvFTD published by the International bvFTD Standards Consortium in 2011;
3. Subjects must not undergo any drug adjustment treatment for 2 months prior to the enrollment and during the enrollment period ;
4. Subjects must sign a written informed consent form prior to the screening visit examination. If the subject cannot sign due to limited cognitive ability or other reasons, the signature may be left blank, and the rationale must be stated. The legal guardian should provide the reason, sign the name, date, and time in the reason description area, and also sign the name, date, and time in the legal guardian column.

Exclusion Criteria:

Inclusion Criteria:

1. Subject is between the ages of 45 - 70;
2. Meetting the diagnostic criteria for "probable bvFTD published by the International bvFTD Standards Consortium in 2011;
3. Subjects must not undergo any drug adjustment treatment for 2 months prior to the enrollment and during the enrollment period ;
4. Subjects must sign a written informed consent form prior to the screening visit examination. If the subject cannot sign due to limited cognitive ability or other reasons, the signature may be left blank, and the rationale must be stated. The legal guardian should provide the reason, sign the name, date, and time in the reason description area, and also sign the name, date, and time in the legal guardian column.

Exclusion Criteria:

1. Dementia caused by other factors: Alzheimer's Disease，vascular dementia, central nervous system infections (such as AIDS, syphilis, etc.), Huntington's disease and Parkinson's disease, Lewy body dementia, traumatic brain injury dementia, other physical and chemical factors (such as drug poisoning, alcohol poisoning, carbon monoxide poisoning, etc.), significant somatic diseases (such as hepatic encephalopathy, pulmonary etc.), intracranial space-occupying lesions (such as subdural hematoma, brain tumors), endocrine system disorders (such as thyroid diseases, parathyroid diseases) and dementia caused by vitamin deficiency or any other known causes;
2. Having a low-carb diet , ketogenic diet, or vegan diet within 3 months before the screening visit or being currently doing.
3. Patients diagnosed with schizophrenia spectrum disorder ,bipolar disorder, moderate to severe depression or delirium according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
4. Abnormal laboratory tests at screening visit and baseline: including liver function tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST]) exceeding twice the upper limit of normal; and renal function (creatinine [Cr]) exceeding 1.5 times the upper limit of normal. Slight exceedances that are not clinically significance, as judged by the investigator, may not be excluded;
5. Fasting triglycerides ≥ 5.7 mmol/L or total cholesterol ≥ 10.34 mmol/L at the screening visit and baseline;
6. Presence any of the following infections at the screening visit:

   Positive human immunodeficiency virus antibody (HIV Ab); Positive Treponema pallidum antibody (TP Ab);
7. Gastrointestinal diseases that could affect the absorption or metabolism of the investigational product as judged by the investigator, within 2 months before the screening visit;
8. Having undergone major surgeries deemed unsuitable for enrollment by the investigator within 6 months before the screening visit or those planning to undergo major surgeries during the study period (The definition of major surgeries refers to Grade 3 and Grade 4 surgeries as outlined in the "Administrative Measures for Grading of Surgeries in Medical Institutions (Trial)" implemented on December 6, 2022);
9. Patients who have suffered from malignant tumors within 3 years prior to the screening visit (excluding basal cell carcinoma of the skin that has been radically cured, squamous cell carcinoma of the skin and/or carcinoma in situ that has been radically resected);
10. Having a history of alcohol or drug abuse within 1 year prior to the screening visit;
11. Known allergy to any components of the investigational product in this study;
12. Having uncorrectable visual or auditory impairments or any other conditions that would affect the assessment of the scale;
13. Contraindications to JT821:

Absolute contraindications:

1. Type 1 diabetes
2. Primary carnitine deficiency (Laboratory tests: Hypoglycemia with low ketone levels, elevated creatine kinase (CK), etc.)
3. Carnitine palmitoyl transferase (CPT) I and II deficiency (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated blood ammonia, tandem mass spectrometry for measurement of blood acylcarnitine profile, etc.)
4. Carnitine translocase deficiency (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated blood ammonia, tandem mass spectrometry for measurement of blood acylcarnitine profile, etc.)
5. β-Oxidation disorders (Laboratory tests: Blood glucose, electrolytes, blood lipids, coagulation, liver function, kidney function)
6. Medium-chain acyl dehydrogenase deficiency (MCAD) (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated blood ammonia, metabolic acidosis, tandem mass spectrometry for measurement of blood acylcarnitine profile, etc.)
7. Very long-chain acyl dehydrogenase deficiency (VLCAD) (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated creatine kinase isoenzyme (CK-MB) and lactate dehydrogenase (LDH), tandem mass spectrometry for measurement of blood acylcarnitine profile)
8. Long-chain acyl dehydrogenase deficiency (LCAD) (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated creatine kinase isoenzyme (CK-MB) and lactate dehydrogenase (LDH), tandem mass spectrometry for measurement of blood acylcarnitine profile)
9. Short-chain acyl dehydrogenase deficiency (SCAD) (Laboratory tests: Tandem mass spectrometry for measurement of blood acylcarnitine profile, determination of SCAD enzyme activity)
10. Long-chain 3-hydroxyacyl-CoA deficiency (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated CK-MB and LDH, analysis of blood acylcarnitine profile, etc.)
11. Medium-chain 3-hydroxyacyl-CoA deficiency (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated CK-MB and LDH, analysis of blood acylcarnitine profile, etc.)
12. Pyruvate carboxylase deficiency (Laboratory tests: Hypoglycemia with low ketone levels, elevated transaminases, CK, elevated CK-MB and LDH, analysis of blood acylcarnitine profile, etc.)
13. Porphyria (Laboratory tests: Sunlight test of urinary porphobilinogen)
14. Acute pancreatitis
15. Liver failure
16. Pregnancy

Relative contraindications:

Patients who cannot maintain adequate nutrition (Fasting blood glucose < 2.8 mmol/L, blood ketone > 0.5 mmol/L) (15) Any other situations that the investigator considers unsuitable for participating in this study; (16)Currently participating in other investigational product/device for treatment or participating in other clinical trials for treatment purposes.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | After 4 and 12 weeks of treatment, changes in MoCa scores relative to baseline.
  After 4 and 12 weeks of treatment, the changes in MoCA scores compared to the baseline MoCA evaluates various cognitive domains including attention, executive functions, memory, language, visuospatial skills, abstraction, calculation, and orientation. It takes about 10 minutes to administer and is scored out of 30 points, with a score of 26 or above considered normal.
Mini-Mental State Examination (MMSE) | After 4 and 12 weeks of treatment, changes in MMSE score relative to baseline.
  After 4 and 12 weeks of treatment, changes in MMSE score compared to the baseline. MMSE tests cognitive function in five areas: orientation, registration, attention and calculation, recall, and language. It consists of 11 questions, with total score ranging from 0-30 points. Lower score indicate greater cognitive impairment.
Clinical Dementia Rating (CDR) scale | After 4 weeks and 12 weeks of treatment, changes relative to baseline
  After 4 and 12 weeks of treatment, changes in CDR score compared to the baseline. CDR assess the progression of dementia, it evaluates six cognitive domains: memory, orientation, judgment/problem solving, community affairs, home and hobbies, and personal care. The CDR provides both a global score and a "Sum of Boxes" score, which ranges from 0 to 18. Higher scores on the CDR indicate more severe dementia.
Frontal Assessment Battery (FAB) | After 4 weeks and 12 weeks of treatment, changes relative to baseline
  After 4 and 12 weeks of treatment, changes in FAB score compared to the baseline. FAB assess frontal lobe functions, with tasks evaluating conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy. The total maximum score is 18, with higher scores indicating better performance.
Neuropsychiatric Inventory (NPI) | After 4 weeks and 12 weeks of treatment, changes relative to baseline
  After 4 and 12 weeks of treatment, changes in NPI score compared to the baseline It evaluates 12 domains including delusions, hallucinations, and apathy, with severity rated from 1 to 3 and frequency from 1 to 4. Higher scores indicate more severe symptoms.
Frontal Behavioral Inventory (FBI) | After 4 weeks and 12 weeks of treatment, changes relative to baseline
  After 4 and 12 weeks of treatment, changes in FBI score compared to the baseline. The FBI is a 24-item caregiver questionnaire that measures behaviors associated with frontal lobe dysfunction, such as apathy and disinhibition. It uses a four-point scale for each item and is scored based on caregiver responses, with higher scores indicating greater impairment.
Boston Naming Test (BNT) | After 4 weeks and 12 weeks of treatment, changes relative to baseline
  After 4 and 12 weeks of treatment, changes in BNT score compared to the baseline. BNT score changes from baseline after 4 and 12 weeks of treatment. The BNT is a quantitative measure of confrontation naming ability, consisting of 60 line drawings of objects. It assesses dysnomia and is sensitive in detecting naming difficulties compared to physical object naming.
Verbal Fluency Test (VFT) | After 4 weeks and 12 weeks of treatment, changes relative to baseline
  After 4 and 12 weeks of treatment, changes in VFT score compared to the baseline.The VFT involves generating words within a category or starting with a specific letter within a time limit. It measures executive functions and language use, with fewer words indicating potential cognitive deficits.

SECONDARY OUTCOMES:
Comparison of the variations in blood ketone values relative to baseline during the treatment period | During the 12-week treatment course
  This measure compares the variations in blood ketone levels relative to the baseline during the treatment period. It also examines the influence of blood ketone levels on cognitive function; higher blood ketone levels are associated with improved cognitive function and therapeutic efficacy.

IPD SHARING:
Plan to Share IPD: No